CLINICAL TRIAL: NCT07215403
Title: Open-Label, Multi-Stage Study to Optimize the Intraputaminal Administration of AB-1005 Using a Prescriptive Infusion Algorithm (PIA)
Brief Title: Prescriptive Infusion Algorithm (PIA)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASK-PD5-CS202
Record Dates: First submitted 2025-09-26; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: PD; Parkinsons Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stage 1 (Experimental): Stage 1 is aimed at evaluating the suitability of PIA-based infusion for standardized intraputaminal administration of AB-1005 via CED under iMRI monitoring.
  Interventions: Procedure: Prescriptive Infusion Algorithm; Drug: AB-1005

INTERVENTIONS:
Procedure: Prescriptive Infusion Algorithm — The study intervention is comprised of the neurosurgical procedure and the bilateral intraputaminal delivery of AB-1005.
Drug: AB-1005 — bilateral intraputaminal delivery of AB-1005

SUMMARY:
This study is being done to test a new way of delivering AB-1005 into the brain. The goal is to make the procedure easier and quicker to perform, while providing similar amounts of drug to the part of the brain that needs treatment.

Technical (Stage 1) To test if the new delivery method (PIA-based infusion) can consistently deliver AB-1005 to the putamen using brain imaging by MRI.

Technical (Stage 2) To confirm the new delivery method works without brain imaging by MRI, using standard operating room tools including brain imaging by CT.

Safety (Stage 1 and 2) To assess the safety and tolerability of the new delivery method for AB-1005 up to 6 months after surgery

DETAILED DESCRIPTION:
Participants will receive a one-time infusion of AB-1005 directly into the putamen on each side of the brain. This is done during a surgical procedure under general anesthesia. The drug is delivered using a special technique called convection-enhanced delivery (CED), which helps spread the drug evenly in the target brain tissue. The delivery method will use either MRI or CT scans to guide and check the placement of the infusion needle (cannula, which is a thin tube).

The study has two main stages, each with two small groups (sub-stages) of 3 participants. Each group will receive the same treatment, and results will be reviewed before moving to the next group.

All participants will receive AB-1005. The study is open-label, meaning both participants and doctors know what treatment is given.

After the follow-up period, all participants will continue into a long-term follow-up (LTFU) study. In the LTFU study, participants' health will be monitored for up to 10 years after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 45 to 75 years of age inclusive, at the time of signing the informed consent.
* >10 years since diagnosis of PD (at time of consenting / Screening Visit 1)
* Presence of bradykinesia plus any of the following:
* Rigidity
* Resting tremor
* Postural instability
* Modified Hoehn and Yahr stage III-IV in the practically defined OFF state
* Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score >40 in the practically defined OFF state
* Stable anti-PD medication regimen for at least 4 weeks prior to Screening Visit 1 and through Baseline Visit
* ≥30% reduction in MDS-UPDRS Part III following a levodopa challenge
* Must agree to use barrier method protection when engaging in intercourse/sexual activity with another person for at least 3 months post-dosing.
* Male participants must refrain from donating sperm for at least 3 months post-dosing.
* Female participants cannot be pregnant or breastfeeding at the time of screening. A woman of childbearing potential (WOCBP) must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) at the required assessments
* Provision of signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Provision of signed consent to also participate in LTFU study ASK-PD0-CS002

Exclusion Criteria:

* Evidence of secondary or atypical parkinsonism (as determined by the neurologist)
* Presence or history of psychosis or impulse control disorder (as determined by the neurologist)
* Presence or history (within 2 years prior to screening) of substance use disorder (including alcohol) as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria (or in the judgment of the neurologist)
* Presence of untreated or sub optimally treated depression (Beck Depression Inventory [BDI]-II score ≥20)
* Current suicidal ideation as indicated by positive response to items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C SSRS), or any history of a suicide attempt
* Clinically significant cognitive impairment (Montreal Cognitive Assessment [MoCA] score <25)
* Presence or history of malignancy other than treated cutaneous squamous or basal cell carcinomas
* Presence of clinically active infection, including acute or chronic scalp infection
* Known contraindications to MRI
* Presence or history of significant cerebrovascular or cardiovascular disease, including:
* Stroke, transient ischemic attack, or other suspected cerebrovascular accident within 1 year prior to screening
* Unstable angina pectoris or myocardial infarction within 1 year prior to screening
* Revascularization procedure(s) within 1 year prior to screening
* Poorly controlled hypertension, poorly controlled diabetes mellitus or prediabetes mellitus with known significant microvascular injury, or other significant cardiovascular history or risk factor
* Known history of complications of anesthesia including difficult airway management and/or difficult endotracheal intubation, malignant hyperthermia, or other related issues that would compromise participant safety during general anesthesia (as determined by the anesthesiologist)
* Inability to identify a safe trajectory to each putamen via an occipitoparietal entry point, or known contraindications to brain surgery in prone position (as determined by the neurosurgeon)
* Known allergy or sensitivity to ingredients in the intervention formulation and/or to gadolinium-based contrast agents
* Concurrent use of percutaneous levodopa/carbidopa intestinal gel, subcutaneous levodopa, or apomorphine pump
* History of brain surgery (including deep brain stimulation [DBS] or focused ultrasound)
* Chronic immunosuppressive therapy
* History of prior cell or gene therapy
* Participation in other interventional clinical trials within 12 weeks prior to screening or unwilling to refrain from starting new investigational agents throughout the course of the study
* Laboratory values at screening:
* Platelets ≤100,000/mm3
* PT >15 s, aPTT >40 s, and/or INR >1.3
* Absolute neutrophil count (ANC) ≤1500/mm3
* Hemoglobin ≤10.0 g/dL
* Aspartate aminotransferase or alanine aminotransferase ≥2.5 times the upper limit of normal
* Total bilirubin ≥2.5 mg/dL
* eGFR <45 mL/min/1.73 m2
* HbA1C ≥8%
* Unable to comply with the protocol procedures, including frequent and prolonged follow-up assessments (during LTFU study ASK-PD0-CS002)
* Unwilling to defer any vaccination from screening through 1 month after surgery
* Any significant issue raised by the neurologist, neurosurgeon, or anesthesiologist that may make a participant unsuitable for the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Amount of the putamen covered by the drug at the end of infusion, assessed by MRI | immediately after the intervention/procedure/surgery
  Investigate the use of PIA-based infusion for consistent intraputaminal administration of AB-1005 via CED under iMRI monitoring

SECONDARY OUTCOMES:
Duration of surgical procedure | through study completion, an average of 1 year
  Reduce the time the surgical procedure is performed
Change in total volumetric putaminal coverage within approximately 60-120 min from end of infusion | immediately after the intervention/procedure/surgery
Accuracy of cannula tip placement at targeted first and last infusion stops in putamen | immediately after the intervention/procedure/surgery

IPD SHARING:
Plan to Share IPD: No